CLINICAL TRIAL: NCT04407780
Title: Cardio-Oncologie: étude Pilote évaluant la faisabilité, Utilité Concrète, Interdisciplinaire d'Une Unité Spécialisée
Brief Title: Cardio-Oncology Registry
Acronym: CONFUCIUS
Status: Recruiting | Type: Observational
Sponsor: European Georges Pompidou Hospital (Other)
Responsible Party: Principal Investigator, Mariana Mirabel, MD, PhD, Assosiate Professor, European Georges Pompidou Hospital
Other Study IDs: 00011928
Record Dates: First submitted 2020-05-14; First posted 2020-05-29 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Cancer; Cardiac Disease; Metabolic Syndrome; Arrhythmia; Heart Diseases
Keywords: cancer; heart; cardiovascular; cardio-oncology; onco-cardiology; phamacology; precision medicine
MeSH Terms: conditions — Neoplasms; Heart Diseases; Metabolic Syndrome; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No interventions are planned — Non applicable

SUMMARY:
Cardio-oncology is an emerging field. Most of the data available have been issued from either retrospective analysis, industry data or pharmacovigilance data. These data sources include a number of bias.

CONFUCIUS is a single tertiary centre prospective registry including all patients who have been referred for cardio-oncology assessemnt.

The objectives are to provide a comprehensive vue of cardoi-oncology, enable to detect early signals of cardiotoxicity and enhance ancillary projetcts aiming at specific populations (e.g., type of cancer) and/or drugs.

ELIGIBILITY:
Inclusion Criteria:

* referred to cardio-oncology

Exclusion Criteria:

* refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All prosepctive patients seen in the cardio-oncology clinic. Observational data will be collected from the medical records. Outcomes measures according to scheduled follow-up visits for their cardiovascular health.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of cardio-toxicty | 5 years
  Number of patients with cardiotoxicity in a cohort of patients referred to a cardio-oncology clinic

SECONDARY OUTCOMES:
Analysis of cardiotoxicity | 5 years
  Correlation of cardio-toxicity overall, and in predefined subgroups; statistical associatoin with outcomes.
Analysis of cardioprotective strategies | 5 years
  Correlation between the use of cardiovascular drugs and the number of patients with cardiotoxicity.
Analysis of underlying cardiovacsular profile | 5 years
  Correlation between underlying cardioascular profile and the number of patients with cardiotoxicity.
Analysis of arrhythmias | 5 years
  Correlation between incident arrhythmias and cancer drugs
Precision medicine | 5 years
  Correlation between biomarkers with use of artificial intelligence and the number of patients with cardiotoxicity.
Oncology | 5 years
  Adherence to oncology treatment plan as stated in the multidisciplinary team meeting in patients with cardio-oncology assessment compared to matched patients with no cardio-oncology assessment within our institution; outcomes.
Cardiovascular outcomes | 10 years
  Assess cardiovascular outcomes (cardiovascular death, admission for heart failure, acute coronary syndrome, stroke).
Any advserse event | 5 years
  Correlation between any adverse event, oncology treatment, and outcomes.
Behaviour | 5 years
  Correlation of any behaviour treatment (exercice, rehabilitation, nutrition consultation) and the number of patents with cardiotoxocity.
Metabolic | 5 years
  Correlation between oncology treatments, cardiovascular therapies, behaviour therapies and the number of patients with metabolic disorders (diabetes or dyslipidemia).

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hôpitaux de Paris - Centre Université de Paris, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Hospital website — http://hopital-georgespompidou.aphp.fr/cardio-oncologie-prevention-cardiovasculaire-2/
- See also: Assistance Publique Hôpitaux de Paris' webinar — https://www.youtube.com/watch?v=_rCgdACAhUU